CLINICAL TRIAL: NCT04035902
Title: Intraoperative IV Iron on the Postoperative Recovery of Red Blood Cell in Hip Arthroplasty Surgery
Brief Title: Intraoperative IV Iron on Postoperative Red Blood Cell Recovery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH 2019-05-008
Record Dates: First submitted 2019-07-21; First posted 2019-07-29 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis, Hip
Keywords: iron; arthroplasty; red blood cell
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ferric carboxymaltose 1000 mg (Experimental): Ferric carboxymaltose is administered during surgery
  Interventions: Drug: Ferric carboxymaltose
- control (Active Comparator): Ferric carboxymaltose is not administered
  Interventions: Drug: control

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferric carboxymaltose is administered during surgery
  Arms: ferric carboxymaltose 1000 mg
Drug: control — Ferric carboxymaltose is not administered
  Arms: control

SUMMARY:
The objective of the present study is to determine the impact of intraoperative IV-iron supplementation on postoperative recovery of RBC mass by retrospectively analyzing and comparing the changes of postoperative hematocrit values after the surgery in patients underwent elective uni-limb total knee arthroplasty surgery with or without IV-iron supplementation during surgery

ELIGIBILITY:
Inclusion criteria

* Patients with osteoarthritis in knee joint undergoing elective uni-limb total knee arthroplasty surgery
* Patients provided a written informed consent.
* Patients with s-ferritin < 300 mg/dl (male) or 200 mg/dl (female)
* Patients with preoperative serum hemoglobin concentration >10 g/dL

Exclusion criteria

* Patients with history of anaphylaxis, iron overload, active infection.
* Patients received or receiving intraoperative and preoperative blood salvaged, allogenic blood transfusion, recombinant human erythropoietin, or undergoing acute normovolemic hemodilution.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
postoperative hematocrit (%) | 7 days after surgery
  hematocrit is evaluated on postoperative 7 days

SECONDARY OUTCOMES:
volume of post-operative bleeding (ml) | 7 day
  total volume of postoperative bleeding collected in the drainage container (hemovac)
intraoperative blood transfusion (ml) | 1 day
  total volume of intraoperative blood transfusion
post-operative blood transfusion (ml) | 7 days
  total amount of post-operative blood transfusion (ml)
post-operative serum ferritin level (ng/ml) | 1 day
  post-operative serum ferritin level (ng/ml) is checked immediately after surgery

IPD SHARING:
Plan to Share IPD: Undecided